CLINICAL TRIAL: NCT02377869
Title: Heavy Light Chain in Chronic Lymphocytic Leukemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Collaborators: Rambam Health Care Campus (Other); Laniado Hospital (Other); Meir Medical Center (Other); Rabin Medical Center (Other); Kaplan Medical Center (Other); Shaare Zedek Medical Center (Other); Hadassah Medical Organization (Other); HaEmek Medical Center, Israel (Other); Western Galilee Hospital-Nahariya (Other Government); Tel-Aviv Sourasky Medical Center (Other Government); Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, tamar.tadmor, MD, Bnai Zion Medical Center
Other Study IDs: 0018-14-BNZ
Record Dates: First submitted 2015-02-25; First posted 2015-03-04 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-02

CONDITIONS: CLL

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervantion

SUMMARY:
Recently, a novel assay for detecting heavy/light chain (HLC) ratios has been reported which enables improvement in paraprotein detection and monitoring in multiple myeloma and other plasma-cell dyscrasias.

The prognostic and biological role of the HLC assay has as yet not been studied in CLL.

Aims of the proposed study:

1. To quantify and analyze the prognostic significance of HLC ratios in the serum of CLL patients. (In addition to FLC)
2. To study the different patterns of Immunoglobulin's subclass antibodies in the serum of patients with CLL and compare them to those of to healthy volunteers.
3. To perform a sub-analysis in patients with CLL who have autoimmune phenomenon (AIHA and ITP)

DETAILED DESCRIPTION:
Analysis of immunoglobulin heavy/light chain pairs In chronic lymphocytic leukemia

Introduction and Background:

Chronic Lymphocytic Leukemia (CLL) is the most common type of leukemia in the western world. Median age at diagnosis is 72 years, and the male to female ratio is 2:1. The disease is characterized by an accumulation of monoclonal mature B-cells which co-express the T-cell antigen CD5, B-cell surface antigens CD19, CD20, and CD23(1) and either kappa or lambda immunoglobulin light chains restriction (2). Diagnosis is established based on the IWCLL criteria published by Hallek at al in 2008. (1).

CLL may have a heterogeneous clinical course with a wide spectrum of manifestations ranging from long lived asymptomatic patients who never require treatment to those with a more rapid clinical course and symptomatic progression. One of the remaining important challenges in CLL is to stratify patients into different prognostic categories, so as to plan appropriate targeted therapy when necessary . The most important prognostic factor in CLL relates to the presence of typical genomic aberrations in the leukemic cell (3). Other essential prognostic parameters include: CD38 expression, the presence of ZAP-70, immunoglobulin heavy chain mutational status, and beta 2 microglobulin (B2MG) levels. (1).

Patients with CLL, have a 10 % risk of developing autoimmune complications mostly auto-immune hemolytic anemia (AIHA) and immune thrombocytopenia (ITP) (4-6). The pathogenesis for these autoimmune cytopenias is linked to the production of polyclonal immunoglobulin G (IgG) antibodies (less frequently IgM) directed against a variety of red blood cell or platelet antigens. (4-6).

The use of serum free light chain (FLC) levels as an important prognostic tool in different plasma cell dyscrasias is already well established (75) while the prognostic significance of FLC in CLL has only been reported more recently by few publications (8-10). Furthermore, Tsai et al, have also described that serum FLC abnormalities may precede diagnosis in 38 % of patients with CLL (11).

Recently, a novel assay for detecting heavy/light chain (HLC) ratios has been reported which enables improvement in paraprotein detection and monitoring in multiple myeloma and other plasma-cell dyscrasias. (12-13).

The prognostic and biological role of the HLC assay has as yet not been studied in CLL.

Aims of the proposed study:

1. To quantify and analyze the prognostic significance of HLC ratios in the serum of CLL patients. (In addition to FLC)
2. To study the different patterns of Immunoglobulin's subclass antibodies in the serum of patients with CLL and compare them to those of to healthy volunteers.
3. To perform a sub-analysis in patients with CLL who have autoimmune phenomenon (AIHA and ITP)

Materials and methods:

The study will be performed in collaboration with the Israeli CLL Study Group.

All patients included will have complete clinical database available and medical records summarized.

Baseline laboratory parameters to be examined will include: complete blood count, Coombs test, serum B2MG and LDH, Immunoglobulin levels,, flow-cytometry including CD38 expression and ZAP70 and urine Bence Jones protein.

Frozen serum samples from CLL patients will be analyzed for levels of:

* Free light chain: kappa/lambda, ratio of K/L and total sum of K+L.
* IgG1, IgG2, IgG3, IgG4.
* Isoforms of heavy/light chain of IgG kappa, IgG lambda, IgA kappa, IgA lambda, IgM kappa, IgM lambda

References:

1. Michael Hallek, Bruce D. Cheson, Daniel Catovsky, et al. Guidelines for the diagnosis and treatment of chronic lymphocytic leukemia: a report from the International Workshop on Chronic Lymphocytic Leukemia updating the National Cancer Institute-Working Group 1996 guidelines. Blood. Jun 15, 2008; 111(12): 5446-5456.
2. Moreau EJ, Matutes E, A'Hern RP, et al. Improvement of the chronic lymphocytic leukemia scoring system with the monoclonal antibody SN8 (CD79b). Am J Clin Pathol.1997;108:378-382.
3. Döhner H, Stilgenbauer S, Benner A, et al. Genomic aberrations and survival in chronic lymphocytic leukemia. N Engl J Med. 2000 Dec 28; 343(26):1910-6.
4. Hamblin TJ, Oscier DG, Young BJ. Autoimmunity in chronic lymphocytic leukemia. J Clin Pathol 1986;39;713-16
5. Zent CS, Kay NE. Autoimmune complications in chronic lymphocytic leukaemia (CLL). Best Pract Res Clin Haematol. 2010 Mar;23(1):47-59.
6. Visco C, Barcellini W, Maura F, Neri A, Cortelezzi A, Rodeghiero F. Autoimmune cytopenias in chronic lymphocytic leukemia. Am J Hematol. 2014 Jun 10
7. Dispenzieri A, Kyle R, Merlini G, et al. International Myeloma Working Group guidelines for serum-free light chain analysis in multiple myeloma and related disorders. Leukemia. 2009 Feb;23(2):215-24.
8. Maurer MJ, Cerhan JR, Katzmann JA, et al. Monoclonal and polyclonal serum free light chains and clinical outcome in chronic lymphocytic leukemia. Blood. 2011 Sep 8;118(10):2821-6
9. Morabito F, De Filippi R, Laurenti L, et al. The cumulative amount of serum-free light chain is a strong prognosticator in chronic lymphocytic leukemia. Blood. 2011 Dec 8;118(24):6353-61.
10. Sarris K, Maltezas D, Koulieris E, et al. Prognostic significance of serum free light chains in chronic lymphocytic leukemia. Adv Hematol. 2013;2013:359071
11. Tsai HT, Caporaso NE, Kyle RA, et al. Evidence of serum immunoglobulin abnormalities up to 9.8 years before diagnosis of chronic lymphocytic leukemia: a prospective study. Blood. 2009 Dec 3;114(24):4928-32
12. Ludwig H, Milosavljevic D, Zojer N, et al. Immunoglobulin heavy/light chain ratios improve paraprotein detection and monitoring, identify residual disease and correlate with survival in multiple myeloma patients. Leukemia. 2013 Apr;27(4):996.
13. Katzmann JA, Clark R, Kyle RA, et al. Suppression of uninvolved immunoglobulins defined by heavy/light chain pair suppression is a risk factor for progression of MGUS. Leukemia. 2013 Jan;27(1):208-12.

ELIGIBILITY:
Inclusion Criteria:

New diagnosed patients with CLL (untreated)

Exclusion Criteria:

Not treated with immunoglobulin Not treated with steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Age>18 years Patients diagnosed with CLL
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
1) To quantify and analyze the prognostic significance of HLC ratios in the serum of CLL patients. (In addition to FLC) | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel, Israel